CLINICAL TRIAL: NCT01994096
Title: Pharmacokinetics and Optimal Dosage of Caspofungin in Critically Ill Patients With Suspected Invasive Candidiasis
Brief Title: Optimal Dosage of Caspofungin in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JWC Alffenaar, PharmD, PhD, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL41676.042.12
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Critically Ill; Suspected Invasive Candidiasis
MeSH Terms: conditions — Critical Illness | interventions — Caspofungin

ARMS (1):
- Caspofungin (Experimental): 1 arm, dose adjustment of caspofungin when exposure is inadequate
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin

SUMMARY:
Intensive care unit (ICU) patients are especially at risk for invasive candidiasis due to the presence of risk factors. It is known that in critically ill patients, alterations in function of various organs and body systems can influence the pharmacokinetics and hence the plasma concentration of a drug. A study of caspofungin in ICU patients has found a high inter- and intra-individual variability in caspofungin concentration. Factors that caused subtherapeutic caspofungin plasma concentrations were body weight > 75 kg and hypoalbuminemia. Furthermore, an efficacy study showed a lower response rate for caspofungin among patients with a higher disease severity score.

As a result of the altered pharmacokinetics, under- or over-exposure of caspofungin can occur in critically ill patients and an adjusted dosage might be necessary in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with caspofungin.
* Admission to an ICU.
* Age ≥ 18 years.
* Suspected invasive candidiasis, established by the physician.

Exclusion Criteria:

* Blood sampling by central venous catheter or peripheral cannula not possible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The optimal dosage of caspofungin in relation to adequate exposure (measured as AUC) in critically ill patients. | 7 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters of caspofungin in critically ill patients. | 3 days
Correlation of pharmacokinetic parameters and the plasma concentration of caspofungin with disease severity scores. | 3 days
Correlation of the plasma concentration of caspofungin with candida eradication. | 28 days
Correlation of the plasma concentration of caspofungin with inflammation parameters. | 3 days
AUC/MIC ratio and highest observed plasma concentration (Cmax)/MIC ratio. | 7 days
Constructing a pharmacokinetic model of caspofungin in critically ill patients. | 28 days
Drug-related adverse events of caspofungin. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, PharmD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] van der Elst KC, Veringa A, Zijlstra JG, Beishuizen A, Klont R, Brummelhuis-Visser P, Uges DR, Touw DJ, Kosterink JG, van der Werf TS, Alffenaar JC. Low Caspofungin Exposure in Patients in Intensive Care Units. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01582-16. doi: 10.1128/AAC.01582-16. Print 2017 Feb. PMID 27855112